CLINICAL TRIAL: NCT06624020
Title: Characteristics and Real-world Use of Palbociclib and Other CDK4/6is in Naive Patients in Australia: a Retrospective Analysis (ROSIE)
Brief Title: A Study to Learn About How Medicines Called CDK4/6 Inhibitors Are Used in People With Advanced or Metastatic Breast Cancer in Australia
Acronym: ROSIE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481187; ROSIE (Other: Alias Study Number)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Breast Cancer Patients: HR+/HER2- metastatic breast cancer patients in in Australia

SUMMARY:
The purpose of this study is to learn about how a class of medicines called CDK4/6 inhibitors, are used for the treatment of breast cancer in patients in Australia. The study looks at how the CDK4/6 inhibitor class of drugs are used for treating breast cancer that is advanced or metastatic (has spread to other parts of the body).

This study does not include patients. Instead, this study looks at already available data to describe characteristics (like age and sex) of patients who have already taken these medicines.

This study will focus on one of these medicines called palbociclib and will look at the data to learn what amounts of the study medicine (palbociclib) patients receive, and how long patients take it for in the real-world in Australia. This study will also learn what other anti-cancer medicines patients receive, including chemotherapy. Chemotherapy is the treatment that uses medicines to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older when first received CDK4/6i breast cancer treatment
* Patient who has received CDK4/6i during study period

Exclusion Criteria:

* There are no exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving CDK4/6i for the first time for HR+ HER2- metastatic breast cancer
Sampling Method: Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Demographic characteristic of participants (CDK4/6i cohort): year of birth | At index date; index date will be defined as the date of dispensation of either any CDK4/6i or palbociclib in the CDK4/6i naive cohort, until Dec 2023
Demographic characteristic of participants (CDK4/6i cohort): sex | At index date; index date will be defined as the date of dispensation of either any CDK4/6i or palbociclib in the CDK4/6i naive cohort, until Dec 2023
Demographic characteristic of participants (CDK4/6i cohort): comorbidities | Within 12 months prior to index date. Index date will be defined as the date of dispensation of either any CDK4/6i or palbociclib in the CDK4/6i naive cohort, until Dec 2023
Demographic characteristic of participants (palbociclib cohort): year of Birth | At index date; index date will be defined as the date of dispensation of either any CDK4/6i or palbociclib in the CDK4/6i naive cohort, until Dec 2023
Demographic characteristic of participants (palbociclib cohort): comorbidities | Within 12 months prior to index date. Index date will be defined as the date of dispensation of either any CDK4/6i or palbociclib in the CDK4/6i naive cohort, until Dec 2023
Demographic characteristic of participants (palbociclib cohort): sex | At index date; index date will be defined as the date of dispensation of either any CDK4/6i or palbociclib in the CDK4/6i naive cohort, until Dec 2023
Proportion of patients receiving palbociclib in combination with aromatase inhibitors or fulvestrant | At index date; Index date will be defined as the date of dispensation of either any CDK4/6i or palbociclib in the CDK4/6i naive cohort, until Dec 2023
Proportion of patients receiving other cancer treatment regimens | At any time from 2004; Within 12 months prior to index date; Within 180 from palbociclib discontinuation until data cut-off, Dec 2023

SECONDARY OUTCOMES:
Treatment continuation rate for palbociclib | At 12 and 24 months from index date until Dec 2023. Index date will be defined as the date of dispensation of either any CDK4/6i or palbociclib in the CDK4/6i naive cohort, until Dec 2023
Percentage of participants with modified doses of palbociclib | First dose modification, from index date until Dec 2023. Index date will be defined as the date of dispensation of either any CDK4/6i or palbociclib in the CDK4/6i naive cohort, until Dec 2023
Median Time to Chemotherapy Initiation from Index | From index date until Dec 2023. Index date will be defined as the date of dispensation of either any CDK4/6i or palbociclib in the CDK4/6i naive cohort, until Dec 2023
Number of comorbidities at initiation of different palbociclib formulations | Within 12 months prior to index date. Index date will be defined as the date of dispensation of either any CDK4/6i or palbociclib in the CDK4/6i naive cohort, until Dec 2023

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Australia, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481187